CLINICAL TRIAL: NCT00241761
Title: Epidemiology of Depression and Heart Failure in Aging
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1312; R01HL079235-04 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure; Heart Failure, Congestive; Depression; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure; Depression; Coronary Disease

SUMMARY:
To understand how depression leads to congestive heart failure (CHF) in older adults.

DETAILED DESCRIPTION:
BACKGROUND:

Depression is known to be associated with an increased risk of coronary heart disease (CHD), and with adverse outcomes among older adults with CHD. Recent evidence suggests that depression is also associated with an increased risk of congestive heart failure, and with adverse outcomes among older adults with congestive heart failure. However, the mechanisms by which depression leads to congestive heart failure are not known

DESIGN NARRATIVE:

To determine the mechanisms of association between depression and CHF, the investigators will use an existing cohort of 1024 older adults (mean age 67) with CHD (including 680 with no heart failure and 344 with clinical or subclinical heart failure) who were recruited between September 2000 and December 2002 for "The Heart and Soul Study." The Heart and Soul Study was originally designed to understand the mechanism of association between depression and CHD. Since patients with CHD are at high risk for CHF, this well-characterized cohort will provide a unique opportunity to examine the relation between depression and CHF. At baseline, participants completed a depression interview (Diagnostic Interview Schedule); full exercise treadmill testing with stress echocardiography; 24-hour Holter monitoring for heart rate variability; 24-hour urine collection for cortisol and norepinephrine; venous blood measurements for lipids, platelet reactivity, and C-reactive protein; and an extensive questionnaire. Participants have been followed annually by telephone. The investigators will invite all participants to return for a 5-year examination, and will follow them for an additional 3 years thereafter, to determine (a) the independent association between baseline depression and CHF, and (b) the extent to which 5-vear changes in biological and behavioral factors associated with depression explain the relation between depression and CHF. By identifying the mechanisms that explain the relation between depression and CHF, this study will enable them to target specific areas for improving the treatment of these patients.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-09; Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Whooley — Northern California Institute for Res & Educ